CLINICAL TRIAL: NCT05177354
Title: Evaluation of Long-term Patient Experience With a Medtronic Closed-Loop Spinal Cord Stimulation System
Brief Title: Medtronic Closed-Loop Spinal Cord Stimulation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT21017
Record Dates: First submitted 2021-11-30; First posted 2022-01-04 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain; Leg Pain; Upper Limb Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Inceptiv

INTERVENTIONS:
Device: Inceptiv — Implantable Neurostimulator with Neuro Sense

SUMMARY:
The purpose of the study is to further understand the closed-loop feature in chronically implanted patients by characterizing the efficacy of the next generation, spinal cord stimulator.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Candidate is undergoing Medtronic SCS device trial for chronic, intractable pain of the trunk and/or limbs
* If being treated for low-back and/or leg pain,

  * the baseline overall^ Visual Analog Scale is ≥ 60 mm and
  * baseline back and/or leg pain Visual Analog Scale is ≥60 mm. ^Average overall pain in the back and/or leg in the 72 hours prior to the baseline visit, measured using Visual Analog Scale.
* If being treated for upper limb pain - baseline Visual Analog Scale is ≥ 60 mm for upper limb pain
* On stable (no change in dose, route, or frequency) prescribed pain medications being used for back and leg pain or upper limb pain, as determined by the investigator, for at least 28 days prior to device trial
* Willing and able to provide signed and dated informed consent
* Willing and able to comply with all study procedures and visits

Exclusion Criteria:

* Indicated for an SCS device to treat stable intractable Angina Pectoris or Peripheral Vascular Disease of Fontaine Stage III or higher
* Previously trialed or implanted with spinal cord stimulator, peripheral or vagus nerve stimulator, deep brain stimulator or an implantable intrathecal drug delivery system
* Currently participating, or plans to participate, in another investigational study unless written approval is provided by the Medtronic study team
* Major psychiatric comorbidity or other progressive diseases that may confound study results, as determined by the Investigator
* Serious drug-related behavioral issues (e.g. alcohol dependency, illegal substance abuse), as determined by the Investigator
* Pregnant or planning on becoming pregnant (if female and sexually active, subject must be using a reliable form of birth control, be surgically sterile, or be at least 2 years post-menopausal)
* Be involved in an injury claim or under current litigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2025-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Russo, MD, Principal Investigator — Genesis Research Services
Locations (7):
- Australia (7):
  - Sydney Pain Specialists, Bella Vista, New South Wales
  - Genesis Research Services, Broadmeadow, New South Wales
  - Australian Medical Research, Hurstville, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Sydney Pain Research Centre, Wahroonga, New South Wales
  - Sunshine Coast Clinical Research, Noosa, Queensland
  - Precision Brain Spine and Pain Center, Kew, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohabbati V, Sullivan R, Yu J, Georgius P, Brooker CD, Siorek M, McClelland NL, Coletti F, Sun X, Franke A, Russo MA. Early outcomes with a flexible ECAP based closed loop using multiplexed spinal cord stimulation waveforms-single-arm study with in-clinic randomized crossover testing. Pain Med. 2025 Nov 1;26(11):773-782. doi: 10.1093/pm/pnaf058. PMID 40378232

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 94 subjects were enrolled. 19 exited prior to the SCS trial. 75 started the trial with 2 subjects not completing the trial and 4 subjects experiencing an unsuccessful trial. Of the 69 that had a successful trial, 9 exited before implant and 60 were implanted. All implanted subjects received SCS therapy following device activation, and subjects with clear and measurable Evoked Compound Action Potentials (ECAPs) had the option to turn the closed loop feature On.
Groups:
- All Implanted Subjects: Enrolled subjects who are implanted with a spinal cord stimulation system. Spinal Cord Stimulation System: Implanted neurostimulation system (neurostimulator and leads) with closed loop feature capabilities.
Period: Implant to 30-day Visit
Arm/Group | All Implanted Subjects
Started | 60
Completed | 57
Not Completed | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lack of compliance to the protocol including phone calls & optimisation visits. | 1
Period: 30-day Visit to 3-Month Visit
Arm/Group | All Implanted Subjects
Started | 57
Completed | 56
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All subjects implanted with a Spinal Cord Stimulator.
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (14.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 47
  More than one race | 10
  Unknown or Not Reported | 0
Primary Location of Pain [Count of Participants; unit: Participants]
  Low-Back and/or Leg Pain | 57
  Upper Limb Pain | 3
Primary Indication [Count of Participants; unit: Participants]
  Degenerative Disk Disease | 23
  Failed Back Syndrome | 20
  Radicular Pain Syndrome | 5
  Post Laminectomy Pain | 4
  Complex Regional Pain Syndrome | 4
  Unsuccessful Disk Surgery | 3
  Peripheral Causalgia | 1
Years Since Onset of Pain [Mean (Standard Deviation); unit: years] | 10.1 (9.69)

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Overstimulation Sensation
Description: The primary outcome is the proportion of low-back and/or leg pain subjects whose average overstimulation intensity score with Closed Loop On is less than their average overstimulation intensity score with Closed Loop Off. During in-clinic testing, subjects perform protocol prescribed activities and rate the intensity of the sensations on a 5-point Likert scale with both Closed Loop On and Off. The average overstimulation intensity scores within each subject are calculated separately for Closed Loop On and Off, and the proportion of subjects with a lower average overstimulation intensity score during Closed Loop On compared to their overstimulation intensity score during Closed Loop Off is calculated with a one-sided 97.5% lower bound.
Time Frame: 30 days from device activation
Population: The pre-specified Primary Analysis Set includes the first 28 low-back and/or leg pain subjects within the All Implanted Subjects Arm with clear and measurable Evoked Compound Action Potentials (ECAPs) who completed in-clinic testing at the 30-day visit. Of the 60 implanted subjects, 2 missed the 30-day visit, 55 completed the 30-day visit, 50 had low-back and/or leg pain and clear and measurable ECAPs, and the first 28 of these subjects are included in the analysis for this objective.
Measure: Count of Participants; unit: Participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 28
Participants | 25
Statistical Analysis 1: Comparison: All Implanted Subjects; Test type: Superiority; p < 0.001, Binomial Exact Test — It is hypothesized that the proportion of low-back and leg pain subjects with a reduction in overstimulation sensation during Closed Loop On compared to Closed Loop Off period exceeds a performance goal of 50%. H0: p ≤ 50% HA: p > 50%; Proportion = 89.3, 97.5% CI 1-sided [lower limit 71.8]

2. Secondary Outcome: Responder Rate for Treatment of Overall Pain
Description: Responder rate defined as a reduction in Overall (back/leg) pain VAS of at least 50%.
Time Frame: 3 months from device activation
Population: All implanted subjects with low-back and/or leg pain who have data at baseline and the 3-month visit. As all subjects were implanted with a spinal cord stimulation system with closed loop feature capabilities, the analysis was pre-specified in the statistical analysis plan to report the combined responder rate for these subjects with data at baseline and the 3-month visit, regardless of whether in-clinic testing of the closed loop feature had been conducted at the 30-day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 51
Participants | 44

3. Secondary Outcome: Responder Rate for Treatment of Low-back Pain
Description: Responder rate defined as a reduction in back pain VAS of at least 50%.
Time Frame: 3 months from device activation
Population: All implanted subjects with low-back pain (baseline VAS ≥ 60mm) who have data at baseline and the 3-month visit. As all subjects were implanted with a spinal cord stimulation system with closed loop feature capabilities, the analysis was pre-specified in the statistical analysis plan to report the combined responder rate for these subjects with data at baseline and the 3-month visit, regardless of whether in-clinic testing of the closed loop feature had been conducted at the 30-day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 43
Participants | 38

4. Secondary Outcome: Responder Rate for Treatment of Leg Pain
Description: Responder rate defined as a reduction in leg pain VAS of at least 50%.
Time Frame: 3 months from device activation
Population: All implanted subjects with leg pain (baseline VAS ≥ 60mm) who have data at baseline and the 3-month visit. As all subjects were implanted with a spinal cord stimulation system with closed loop feature capabilities, the analysis was pre-specified in the statistical analysis plan to report the combined responder rate for these subjects with data at baseline and the 3-month visit, regardless of whether in-clinic testing of the closed loop feature had been conducted at the 30-day visit.
Measure: Count of Participants; unit: Participants
Arm/Group | All Implanted Subjects
Number analyzed (Participants) | 41
Participants | 30

ADVERSE EVENTS:
Time Frame: From Implant through 3 months post activation
Description: All device/therapy-related adverse events (AEs) related to the implanted spinal cord stimulation (SCS) system, accessories, surgical procedures, and therapy were collected. Non-serious, non-device/therapy-related AEs were not collected. All serious AEs were collected regardless of device/therapy-relatedness. AEs were not collected separately by whether the closed loop feature was On or Off; it was pre-specified to report the AE rates through the 3-month visit for all implanted subjects.
Arm/Group | All Implanted Subjects
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 10/60
Other Adverse Events (participants affected / at risk) | 3/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Implanted Subjects (N=60)
Medical device site infection (Infections and infestations) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 1 (1)
Medical device site pain (General disorders) | 1 (1)
Medical device site hematoma (General disorders) | 1 (1)
Staphylococcal bacteremia (Infections and infestations) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1)
Dysponea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Implanted Subjects (N=60)
Medical device site pain (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution must ensure the Discloser gives a copy of any proposed Publication drafted by them and/or Personnel involved in the conduct of the Study to the Sponsor at least 40 days The Sponsor may do one of the following

1. provide optional comments
2. request delay for no more than 120 days to file patent applications or take other measures to preserve or secure its IP, Institution must abide by request
3. request removal of Confidential Information from the Publication

DOCUMENTS (2):
  • Study Protocol (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT05177354/Prot_003.pdf
  • Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT05177354/SAP_004.pdf